CLINICAL TRIAL: NCT03262012
Title: A Randomized, Double-Blind, Parallel-Group, 28-Week, Chronic-Dosing, Multi-Center, Extension Study to Assess the Safety and Efficacy of PT010, PT003, and PT009 in Japanese Subjects With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD) Compared With Symbicort® Turbuhaler® as an Active Control
Brief Title: Study to Assess the Safety and Efficacy of PT010, PT003, and PT009 in Japanese Subjects With COPD Compared With Symbicort® Turbohaler®
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT010007
Record Dates: First submitted 2016-02-17; First posted 2017-08-25 (Actual); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- BGF MDI (PT010) (Experimental): Budesonide, Glycopyrronium, and Formoterol Fumarate Inhalation Aerosol, BGF MDI, PT010
  Interventions: Drug: BGF MDI (PT010)
- GFF MDI (PT003) (Experimental): Glycopyrronium and Formoterol Fumarate Inhalation Aerosol, GFF MDI, PT003
  Interventions: Drug: GFF MDI (PT003)
- BFF MDI (PT009) (Experimental): Budesonide and Formoterol Fumarate Inhalation Aerosol, BFF MDI, PT009
  Interventions: Drug: BFF MDI (PT009)
- Symbicort® Turbohaler® Inhalation Powder (Active Comparator): Budesonide and Formoterol Fumarate Inhalation Powder, Symbicort® Turbohaler® Inhalation Powder, Symbicort Turbohaler
  Interventions: Drug: Symbicort® Turbohaler® Inhalation Powder

INTERVENTIONS:
Drug: BGF MDI (PT010) — Budesonide, Glycopyrronium, and Formoterol Fumarate Inhalation Aerosol, BGF MDI, PT010
  Other Names: BGF
  Arms: BGF MDI (PT010)
Drug: GFF MDI (PT003) — Glycopyrronium and Formoterol Fumarate Inhalation Aerosol, GFF MDI, PT003
  Other Names: GFF
  Arms: GFF MDI (PT003)
Drug: BFF MDI (PT009) — Budesonide and Formoterol Fumarate Inhalation Aerosol, BFF MDI, PT009
  Other Names: BFF
  Arms: BFF MDI (PT009)
Drug: Symbicort® Turbohaler® Inhalation Powder — Budesonide and Formoterol Fumarate Inhalation Powder, Symbicort® Turbohaler® Inhalation Powder, Symbicort Turbohaler
  Other Names: Symbicort
  Arms: Symbicort® Turbohaler® Inhalation Powder

SUMMARY:
A Randomized, Double-Blind, Parallel Group, 28-Week Chronic Dosing, Multi-Center Long-term Extension Study to Assess the Safety and Efficacy in Japanese Subjects with Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD) compared with Symbicort® Turbohaler®

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel group, chronic dosing, active-controlled, 28-week, safety extension of Study PT010006 to assess the safety and efficacy of BGF MDI, GFF MDI, BFF MDI, and Symbicort TBH as an active control over a 52-week period in Japanese subjects with moderate to very severe COPD who remain symptomatic on maintenance treatment with either an ICS and one or more bronchodilator(s) or two or more maintenance bronchodilators.

ELIGIBILITY:
Inclusion Criteria

* Given their signed written informed consent to participate.
* Subjects must have agreed to participate and complete the lead-in Study PT010006.
* Non-child bearing potential (ie, physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal); or Child bearing potential, has a negative serum pregnancy test at Visit 1, and agrees to acceptable contraceptive methods used consistently and correctly for the duration of the study.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS), or other local applicable guidelines.
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking.
* Forced expiratory volume in 1 second (FEV1)/Forced vital capacity (FVC) ratio must be <0.70 and FEV1 must be <80% predicted normal value calculated using NHANES III reference equations (or reference norms applicable to other regions).
* Required COPD maintenance therapy:
* All Subjects must have been on two or more inhaled maintenance therapies for the management of their COPD for at least 6 weeks prior to Screening. Scheduled SABA and/or scheduled SAMA are considered inhaled maintenance therapies.

Please refer to the study protocol for the complete inclusion criteria list.

Exclusion Criteria

* Significant diseases or conditions other than COPD, which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
* Women who are pregnant or lactating, or are planning to become pregnant during the course of the study, or women of childbearing potential who are not using an acceptable method of contraception.
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma.
* Subjects who have been hospitalized due to poorly controlled COPD within 3 months prior to Visit 1 (Screening) or during the Screening Period
* Subjects who have poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to Visit 1 (Screening) or during the Screening Period
* Immune suppression or severe neurological disorders affecting control of the upper airway or other risk factors that in the opinion of the Investigator would put the subject at substantial risk of pneumonia.
* Subjects with a diagnosis of narrow angle glaucoma, who, in the opinion of the Investigator, have not been adequately treated.
* Subjects who have a history of hypersensitivity to β2-agonists, budesonide or any other corticosteroid components, glycopyrronium or other muscarinic anticholinergics, or any other component of the IMPs.

Please refer to the study protocol for the complete exclusion criteria list.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M. Dorinsky, MD, Study Director — Pearl Therapeutics, Inc.
Locations (61):
- Japan (61):
  - Research Site, Bunkyō City
  - Research Site, Chūōku
  - Research Site, Date-gun
  - Research Site, Fukuoka
  - Research Site, Ginowan-shi
  - Research Site, Hakata-shi
  - Research Site, Hamamatsu
  - Research Site, Higashiokitama-gun
  - Research Site, Higashiosaka-shi
  - Research Site, Himeji-shi
  - Research Site, Hirakata-shi
  - Research Site, Iizuka-shi
  - Research Site, Itabashi-ku
  - Research Site, Iwata-shi
  - Research Site, Izumo-shi
  - Research Site, Kagoshima
  - Research Site, Kahoku-gun
  - Research Site, Kakogawa-shi
  - Research Site, Kasaoka-shi
  - Research Site, Kasuga-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kiyose-shi
  - Research Site, Kobe
  - Research Site, Koga-shi
  - Research Site, Kurashiki-shi
  - Research Site, Kure-shi
  - Research Site, Kyoto
  - Research Site, Maebashi
  - Research Site, Matsumoto-shi
  - Research Site, Matsusaka-shi
  - Research Site, Meguro-ku
  - Research Site, Mitaka-shi
  - Research Site, Mizunami-shi
  - Research Site, Nagaoka-shi
  - Research Site, Nagoya
  - Research Site, Naha
  - Research Site, Nishishirakawa-gun
  - Research Site, Obihiro-shi
  - Research Site, Ogaki-shi
  - Research Site, Okinawa-shi
  - Research Site, Ookawa-shi
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Ōita
  - Research Site, Ōtsu
  - Research Site, Sakaide-shi
  - Research Site, Sakaishi
  - Research Site, Sapporo
  - Research Site, Sendai
  - Research Site, Seto-shi
  - Research Site, Shinagawa-ku
  - Research Site, Shinjuku-ku
  - Research Site, Shizuoka
  - Research Site, Suita-shi
  - Research Site, Tachikawa-shi
  - Research Site, Takamatsu
  - Research Site, Toon-shi
  - Research Site, Toshima-ku
  - Research Site, Toyama
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Singh D, Hurst JR, Martinez FJ, Rabe KF, Bafadhel M, Jenkins M, Salazar D, Dorinsky P, Darken P. Predictive modeling of COPD exacerbation rates using baseline risk factors. Ther Adv Respir Dis. 2022 Jan-Dec;16:17534666221107314. doi: 10.1177/17534666221107314. PMID 35815359

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 75 study centers in Japan, from Aug 2016 to June 2018. This is an extension study of PT010006 and could take up to an additional 28 weeks.
Pre-assignment Details: Subjects were randomized in a 2:2:1:1 scheme.
Groups:
- BGF MDI 320/14.4/9.6 ug: Budesonide Gylcopyrronium and Formoterol Fumarate Inhalation Aerosol 320/14.4/9.6 ug
- GFF MDI 14.4/9.6 ug: Glycopyrronium and Formoterol Fumarate Inhalation Aerosol 14.4/9.6 ug
- BFF MDI 320/9.6 ug: Budesonide and Formoterol Fumarate Inhalation Aerosol 320/9.6 ug
- Symbicort TBH 400/12 ug BID: Open Label Symbicort Turbuhaler 400/12 ug BID
Period: Overall Study
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug | Symbicort TBH 400/12 ug BID
Started | 139 | 138 | 70 | 69
Completed | 112 | 102 | 56 | 54
Not Completed | 27 | 36 | 14 | 15
Not completed — Withdrawal by Subject | 15 | 13 | 8 | 7
Not completed — Adverse Event | 10 | 12 | 4 | 6
Not completed — Physician Decision | 2 | 5 | 1 | 0
Not completed — Lack of Efficacy | 0 | 5 | 1 | 2
Not completed — Protocol Discontinuation Criteria | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Japanese Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug | Symbicort TBH 400/12 ug BID | Total
Number analyzed (Participants) | 139 | 138 | 70 | 69 | 416
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Japanese Safety Population
  Years | 69.4 (7.1) | 69.0 (6.1) | 69.7 (6.1) | 70.1 (6.8) | 69.5 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Japanese Safety Population
  Participants
    Female | 9 | 12 | 2 | 1 | 24
    Male | 130 | 126 | 68 | 68 | 392
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Japanese subjects randomized
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 139 | 138 | 69 | 69 | 415
    Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Japanese subjects randomized
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 139 | 138 | 70 | 69 | 416
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Post-baseline Newly Occurring or Worsening PCS (Potentially Clinically Significant) Clinical Chemistry Values
Description: Number of participants post-baseline newly occurring or worsening PCS (potentially clinically significant) clinical chemistry values
Time Frame: 28 Weeks
Population: Japanese Safety Population
Measure: Number; unit: Count of Participants
Groups:
- Symbicort TBH 400/12 ug: Open Label Symbicort Turbuhaler 400/12 ug BID
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug | Symbicort TBH 400/12 ug
Number analyzed (Participants) | 137 | 137 | 68 | 68
Count of Participants
  ALT >3 x ULN | 0 | 1 | 0 | 0
  Total Bilirubin >2 x ULN | 0 | 0 | 0 | 1
  Potassium (mmol/L) >6.0 | 2 | 0 | 0 | 0
  Glucose (mmol/L) >13.9 if Baseline is ≤10.0 | 0 | 1 | 1 | 1
  Glucose (mmol/L) >16.7 if baseline is >10.0 | 0 | 1 | 0 | 0

2. Primary Outcome: Incidence of Post-baseline Newly Occurring or Worsening PCS Vital Signs
Description: Incidence of Post-baseline Newly Occurring or Worsening PCS Vital Signs
Time Frame: 28 Weeks
Population: Japanese Safety Population
Measure: Number; unit: Particpants
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug | Symbicort TBH 400/12 ug
Number analyzed (Participants) | 139 | 138 | 70 | 69
Particpants
  Systolic Blood Pressure >=180, Incr >=20 | 3 | 1 | 0 | 0
  Systolic Blood Pressure, <=90, Decr >=20 | 4 | 1 | 1 | 1
  Diastolic Blood Pressure, >=105 Incr, >=15 | 2 | 1 | 2 | 0
  Diastolic Blood Pressure, <=50, Decr >=15 | 4 | 3 | 2 | 3
  Tachycardia Event >=110, Incr >=15% | 1 | 0 | 2 | 0
  Bradycardia Event <=50, Decr >=15% | 9 | 8 | 3 | 2

3. Primary Outcome: Incidence of Post-baseline Newly Occurring or Worsening PCS ECG Values
Description: Incidence of Post-baseline Newly Occurring or Worsening PCS ECG Values
Time Frame: 28 Weeks
Population: Japanese Safety Population
Measure: Number; unit: Participants
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug | Symbicort TBH 400/12 ug
Number analyzed (Participants) | 139 | 138 | 70 | 69
Participants
  >=500 if <500 msec at BL and change >=15 msec | 1 | 0 | 0 | 0
  >=530 if >=500 msec at BL and >=15 msec | 0 | 0 | 0 | 0
  >= 500 msec and >= 15 msec change from BL | 1 | 0 | 0 | 0
  Increase from baseline is >=60 msec | 1 | 1 | 0 | 0
  Value is >500 msec and increase >=60 msec | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed informed consent throughout the treatment period and up to 14 days following the last dose of study drug up to an average of 30 weeks.
Description: The Study safety population was defined as all subjects who signed ICF for PT010006 and received any amount of study treatment.
Arm/Group | BGF MDI 320/14.4/9.6 ug | GFF MDI 14.4/9.6 ug | BFF MDI 320/9.6 ug | Symbicort TBH 400/12 ug BID
All-Cause Mortality (participants affected / at risk) | 3/139 | 1/138 | 1/70 | 1/69
Serious Adverse Events (participants affected / at risk) | 21/139 | 30/138 | 11/70 | 14/69
Other Adverse Events (participants affected / at risk) | 82/139 | 75/138 | 40/70 | 38/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI 320/14.4/9.6 ug (N=139) | GFF MDI 14.4/9.6 ug (N=138) | BFF MDI 320/9.6 ug (N=70) | Symbicort TBH 400/12 ug BID (N=69)
Chronic obstructive pulmonary disorder (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 11 (21) | 2 (2) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 3 (3) | 1 (1) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm of thymus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGF MDI 320/14.4/9.6 ug (N=139) | GFF MDI 14.4/9.6 ug (N=138) | BFF MDI 320/9.6 ug (N=70) | Symbicort TBH 400/12 ug BID (N=69)
Nasopharyngitis (Infections and infestations) | 45 (69) | 43 (57) | 22 (33) | 24 (30)
Bronchitis (Infections and infestations) | 14 (20) | 11 (20) | 8 (10) | 7 (8)
Influenza (Infections and infestations) | 5 (5) | 6 (6) | 3 (3) | 6 (6)
Upper Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 5 (8) | 7 (9) | 5 (7) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 1 (1) | 9 (9) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 (16) | 6 (6) | 6 (7) | 3 (3)
Constipation (Gastrointestinal disorders) | 6 (6) | 5 (8) | 4 (4) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 4 (4) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 8 (12) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT03262012/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT03262012/SAP_001.pdf